CLINICAL TRIAL: NCT03464552
Title: Role of Oral Celecoxib 200 mg in Reducing Pain Associated With Colposcopic Directed Biopsy: A Randomized Triple-blind Placebo-controlled Trial
Brief Title: Celecoxib in Colposcopic Directed Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed AA Wali, MD, Lecturer of Obstetrics and Gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-2aa6-2018
Record Dates: First submitted 2018-03-02; First posted 2018-03-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Colposcopy
Keywords: colposcopy - colposcopic directed biopsy - celecoxib
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Celecoxib group (Active Comparator): will receive oral Celecoxib 200 mg capsule (Celebrex®200, Pfizer, USA) once 3 hours before the colposcopic guided biopsy
  Interventions: Drug: Celecoxib 200mg; Procedure: Colposcopic guided biopsy
- Placebo group (Placebo Comparator): will receive oral placebo capsule once 3 hours before the colposcopic guided biopsy
  Interventions: Procedure: Colposcopic guided biopsy; Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Celecoxib 200mg — oral capsule 3 hours before procedure
  Other Names: celebrex 200
  Arms: Celecoxib group
Procedure: Colposcopic guided biopsy — Patient is placed in the lithotomy position. Vulva is examined for any suspicious lesions. A sterile bivalve speculum is introduced into the vagina to inspect cervix. A 3% acetic acid solution is applied to the cervix to map acetowhite areas for colposcopic directed punch biopsy using Tischler punch forceps.
Drug: Placebo oral capsule — oral capsule 3 hours before procedure
  Arms: Placebo group

SUMMARY:
Women often experience pain and discomfort during colposcopic examination especially at time of colposcopic directed excisional biopsy, pre-procedure anxiety, women pain threshold may also increase pain, woman's cooperation during the procedure is affected by all these factors, which also may hinder the colposcopist from obtaining adequate data and biopsies.

Several pharmacological and non-pharmacological methods have been studied to reduce pain associated colposcopic directed biopsy (CDB). We aim to study the effect of Celecoxib to reduce pain associated with CDB.

ELIGIBILITY:
Inclusion Criteria:

• Females 18-65 years old who undergoing colposcopic directed biopsy

Exclusion Criteria:

* A known allergy to Celecoxib, aspirin or another NSAID.
* Active peptic ulceration or gastrointestinal bleeding.
* Inflammatory bowel disease.
* Congestive heart failure (NYHA II-IV).
* Established ischemic heart disease, peripheral arterial disease and/or cerebrovascular disease.
* History of neurologic deficit.
* Known hepatic or renal impairment.
* Pregnancy.
* Breast-feeding.
* Post-hysterectomy.
* Bleeding disorders.
* Drug abuse.
* Cervical and vaginal infection.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 170 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Pain during the procedure | Immediately after the first biopsy
  Visual analog score in mm on a 10 cm ruler

SECONDARY OUTCOMES:
Pain at time of vaginal speculum application | At time of introduction of vaginal speculum
  Visual analog score in mm on a 10 cm ruler
Post-procedure pain | At 30 minutes after completing the procedure
  Visual analog score in mm on a 10 cm ruler

OTHER OUTCOMES:
Effect of pain score on duration of the colposcopic procure | At time of removal of vaginal speculum
  Duration in minutes (from introduction of vaginal speculum till its removal)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided